CLINICAL TRIAL: NCT07040618
Title: Assessing the Effectiveness of Rhomboid Intercostal and Erector Spinae Plane Blocks After Lung Cancer Thoracotomy
Brief Title: Rhomboid Intercostal Block vs Erector Spinae Block
Acronym: RIB-ESPB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sayed Mahmoud Abed, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-CAIRO-RIb-ESPB-2025
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a parallel-group randomized controlled trial comparing the effectiveness of two ultrasound-guided regional anesthesia techniques-Rhomboid Intercostal Block (RIB) and Erector Spinae Plane Block (ESPB)-in managing postoperative pain in lung cancer patients undergoing thoracotomy.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided Rhomboid Intercostal Block (Experimental): Patients in this group will receive a rhomboid intercostal block with 20-25 mL of 0.25% bupivacaine injected between the rhomboid major and intercostal muscles under ultrasound guidance 30-45 minutes before surgery.
  Interventions: Procedure: Ultrasound-guided Rhomboid Intercostal Block
- Ultrasound-guided Erector Spinae Plane Block (Active Comparator): Patients in this group will receive an erector spinae plane block with 20-25 mL of 0.25% bupivacaine injected deep to the erector spinae muscle at the T4-T5 level under ultrasound guidance 30-45 minutes before surgery.
  Interventions: Procedure: Ultrasound-guided Erector Spinae Plane Block

INTERVENTIONS:
Procedure: Ultrasound-guided Rhomboid Intercostal Block — This intervention involves an ultrasound-guided injection of 20-25 mL of 0.25% bupivacaine into the fascial plane between the rhomboid major and intercostal muscles. The patient is positioned laterally, and the block is performed at the T5-T6 level using a high-frequency linear ultrasound probe. The goal is to anesthetize the lateral cutaneous branches of the intercostal nerves to provide postoperative thoracic analgesia.
  Arms: Ultrasound-guided Rhomboid Intercostal Block
Procedure: Ultrasound-guided Erector Spinae Plane Block — This intervention consists of an ultrasound-guided injection of 20-25 mL of 0.25% bupivacaine into the plane deep to the erector spinae muscle at the T4-T5 transverse process level. The patient is positioned sitting or in lateral decubitus, and the procedure uses a curved or linear ultrasound probe. This block targets the dorsal and ventral rami of thoracic spinal nerves to manage postoperative pain after thoracotomy.
  Arms: Ultrasound-guided Erector Spinae Plane Block

SUMMARY:
This randomized trial compares rhomboid intercostal block (RIB) and erector spinae plane block (ESPB) for postoperative pain control in lung cancer patients undergoing thoracotomy. Sixty patients will be assessed for 24-hour morphine consumption, pain scores, hemodynamics, recovery time, satisfaction, and side effects. The study aims to identify the more effective technique for enhancing recovery and minimizing opioid use.

DETAILED DESCRIPTION:
This randomized clinical trial aims to evaluate the analgesic efficacy of two ultrasound-guided regional anesthesia techniques-Rhomboid Intercostal Block (RIB) and Erector Spinae Plane Block (ESPB)-in female lung cancer patients undergoing thoracotomy at the National Cancer Institute, Cairo University. Thoracotomy is known for causing severe postoperative pain, which, if not effectively managed, can lead to chronic pain and impaired pulmonary function. Traditional techniques like thoracic epidural or paravertebral blocks, while effective, have limitations due to technical complexity and potential complications. Recently, interfascial plane blocks such as ESPB have shown promise for thoracic analgesia, and RIB has emerged as a technique potentially offering superior lateral thoracic wall coverage.

Sixty patients will be randomly assigned to receive either RIB or ESPB 30-45 minutes before surgery. The primary outcome is 24-hour postoperative morphine consumption. Secondary outcomes include visual analog scale (VAS) pain scores, hemodynamic stability, time to first analgesic request, recovery duration, patient satisfaction, and incidence of nausea and vomiting.

General anesthesia will be standardized across both groups. Data will be analyzed using appropriate statistical tests, and ethical approval will be obtained prior to patient enrollment. This study supports multimodal analgesia and aims to inform clinical practice in pain management after oncologic thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thoracotomy for lung cancer

Age ≥ 18 years and ≤ 65 years

ASA physical status II or III

Body Mass Index (BMI) > 20 kg/m² and < 35 kg/m²

Willing and able to provide informed consent

Exclusion Criteria:

Patient refusal

ASA physical status IV

Age < 18 years or > 65 years

BMI < 20 kg/m² or > 35 kg/m²

Known allergy or contraindication to local anesthetics or opioids used in the study

History of chronic pain or psychological disorders

Contraindications to regional anesthesia (e.g., local infection, coagulopathy, pre-existing peripheral neuropathy)

Severe respiratory, cardiac, hepatic, or renal disease

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
24-hour postoperative morphine consumption | Within the first 24 hours postoperatively
  This outcome measures the total amount of morphine (in milligrams) administered to each patient within the first 24 hours after thoracotomy. Morphine will be given as rescue analgesia when the patient reports a visual analog scale (VAS) pain score of 4 or more. The cumulative dose will be recorded and compared between the Rhomboid Intercostal Block (RIB) and Erector Spinae Plane Block (ESPB) groups to evaluate the relative effectiveness of each regional anesthesia technique in managing postoperative pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed M Abed, MD, Principal Investigator — Associate Professor of Anesthesia and Pain Management, National Cancer Institute -- Cairo University
Locations (1):
- National Cancer Institute - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to institutional policy and privacy concerns. The study involves sensitive patient data from a cancer population, and data sharing may pose risks to confidentiality despite de-identification efforts. Access will remain restricted to the research team at the National Cancer Institute, Cairo University, in accordance with ethical approval and informed consent protocols.

REFERENCES:
- See also: The morbidity, time course and predictive factors for persistent post-thoracotomy pain — https://pubmed.ncbi.nlm.nih.gov/11394926/
- See also: In patients undergoing thoracic surgery is paravertebral block as effective as epidural analgesia for pain management? — https://pubmed.ncbi.nlm.nih.gov/19854794/